CLINICAL TRIAL: NCT03367377
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3209590 Following Multiple Weekly Doses in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of LY3209590 in Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16392; I8H-MC-BDCB (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-12-05; First posted 2017-12-08 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3209590 (Experimental): Escalating doses of LY3209590 administered by subcutaneous (SC) injection
  Interventions: Drug: LY3209590
- Insulin glargine (Active Comparator): Insulin glargine administered by SC injection
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: LY3209590 — Administered SC
  Arms: LY3209590
Drug: Insulin Glargine — Administered SC
  Arms: Insulin glargine

SUMMARY:
This study will evaluate the safety and tolerability of LY3209590 when given by injection under the skin to participants with type 2 diabetes. It will also investigate how the body processes the study drug and the effect of the study drug on blood sugar levels. Information about any side effects will be documented.

This study will last approximately 17 weeks, not including screening. Screening is required within 4 weeks prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Type 2 Diabetes Mellitus (T2DM) for at least 1 year
* Have a glycated hemoglobin (HbA1c) greater than or equal to (≥) 7.0 percent (%) to less than or equal to (≤) 10.5% at screening
* Have had no episodes of severe hypoglycemia in the past 6 months
* Are on stable basal insulin (neutral protamine Hagedorn insulin suspension [NPH] insulin, insulin glargine [U100 or U300], or insulin detemir) with or without metformin, dipeptidyl peptidase IV (DPP-IV) inhibitors, sulfonylureas, and sodium-glucose co-transporter 2 (SGLT-2) inhibitors, at a stable dose for at least 3 months before screening

Exclusion Criteria:

* Have significant lipohypertrophy in the target abdominal injection
* Have a history of renal impairment
* Have a history of deep vein thrombosis of the leg or repeated episodes of deep leg vein thrombosis in first-degree relatives (parents, siblings, or children)
* Have proliferative retinopathy or maculopathy and/or severe neuropathy
* Any significant changes in insulin regimen and/or unstable blood glucose control within the past 3 months prior to screening
* Require daily insulin treatment less than (<) 0.15 unit/kilogram (U/kg) per body weight
* Are treated with a continuous subcutaneous insulin infusion (CSII) pump
* Currently receiving degludec insulin therapy, or have been treated with degludec within the past 90 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-10-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through 17 weeks
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Drug Plasma Concentration Versus Time Curve from Time Zero to 168 hours (AUC[0-168]) of LY3209590 | Week 6
  PK: AUC(0-168) of LY3209590
Pharmacodynamics (PD): Average Glucose from 7-Point Glucose Profiles | Baseline, Day 4, Day 40, Day 43
  PD: Average Glucose from 7-Point Glucose Profiles

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (2):
  - Miami Research Associates, South Miami, Florida
  - High Point Clinical Trials Center, High Point, North Carolina
- LMC Endocrinology Centres Ltd., Toronto, Ontario, Canada

REFERENCES:
- See also: A Study of LY3209590 in Participants With Type 2 Diabetes — https://www.lillytrialguide.com/en-US/studies/adult-type-2-diabetes/BDCB#?postal=